CLINICAL TRIAL: NCT03186508
Title: Enhancing Sleep Duration: Effects on Children's Eating and Activity Behaviors-Renewal
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Temple University (Other)
Collaborators: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: R01HL092910 (NIH); R01HL092910 (NIH)
Record Dates: First submitted 2017-03-31; First posted 2017-06-14 (Actual); Last update posted 2024-10-28 (Actual); Status verified 2024-01

CONDITIONS: Obesity; Sleep
Keywords: obesity prevention; sleep; behavioral intervention
MeSH Terms: conditions — Obesity

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Optimize Sleep (OS) (Active Comparator): Optimize Sleep will focus exclusively on enhancing sleep by using effective behavioral strategies. Specific strategies to be used include: goal setting and self-monitoring, positive bedtime routines, stimulus control/sleep hygiene strategies, problem-solving regarding challenges, and review of effective strategies for relapse prevention.
  Interventions: Behavioral: Optimize Sleep (OS)
- Optimize Sleep-Plus (OS-Plus) (Active Comparator): OS-Plus will focus on enhancing sleep and targeted eating (decreasing sugar-sweetened beverages and sweet and salty snack foods) and activity (increasing physical activity and decreasing TV viewing) behaviors. Specific strategies to be used include: goal setting and self-monitoring, positive bedtime routines, stimulus control/sleep hygiene strategies, problem-solving regarding challenges, and review of effective strategies for relapse prevention.
  Interventions: Behavioral: Optimize Sleep-Plus (OS-Plus)

INTERVENTIONS:
Behavioral: Optimize Sleep (OS) — All children will receive 8 sessions during active treatment: two in-person weekly, three in-person biweekly, and 3 monthly sessions conducted by phone. All families will be asked to complete 3 "sleep challenges" (at weeks 8, 16, and 20). During maintenance, families will continue with monthly phone contact.
  Arms: Optimize Sleep (OS)
Behavioral: Optimize Sleep-Plus (OS-Plus) — All children will receive 8 sessions during active treatment: two in-person weekly, three in-person biweekly, and 3 monthly sessions conducted by phone. All families will be asked to complete 3 "sleep challenges" (at weeks 8, 16, and 20). During maintenance, families will continue with monthly phone contact.
  Arms: Optimize Sleep-Plus (OS-Plus)

SUMMARY:
Enhancing children's sleep may be a novel approach for prevention of obesity and cardiovascular (CV) disturbance. Observational studies with children demonstrate that short sleep increases risk of obesity and other CV risk factors. Randomized controlled trials with children 8-11 years old demonstrate that enhancing sleep duration leads to positive changes in eating and activity behaviors and weight status, particularly for children who enhance their sleep the most. Enhancing sleep may be particularly important for racial minority children and those from lower socioeconomic backgrounds given their increased risk for short sleep, obesity and CV risk factors. In this study two active obesity preventive interventions will be evaluated: a) enhancing sleep alone (Optimize Sleep [OS]), and b) enhancing sleep along with eating and activity behaviors that have demonstrated efficacy for obesity prevention and are implicated in self-regulatory pathways related to sleep (i.e., energy dense snack foods and beverages, TV viewing, and physical activity) (OS-Plus). Two hundred four children 6-11 years old who are primarily African American/black, primarily from low socioeconomic backgrounds, and who sleep < 9.5 hours/night into a 12-month study will be enrolled. Children will be randomly assigned to either OS or OS-Plus. Over the 6-month treatment phase, all children will attend an 8-session treatment; monthly phone contacts will occur during maintenance (6-12 months). Primary aim is to determine the efficacy of OS-Plus relative to OS on change in body mass index z-score (BMIz) at end of treatment. Secondary aims will assess efficacy of OS-Plus relative to OS on additional cardiometabolic risk factors, eating and activity behaviors. Exploratory aims will assess maintenance of effects at 12 months.

ELIGIBILITY:
Inclusion Criteria:

1. Caregiver-reported child age of 6-11 years
2. < 9.5 Hours time-in-bed for sleep most days/week
3. BMI for age and gender > 25th percentile (but no greater than 100% overweight)
4. Understanding of and ability to complete protocol
5. Self-reported caregiver age of 18 years and primary caregiver at bedtimes/wake times
6. Likes food used in the eating regulation paradigms
7. Willingness to be randomized to either treatment condition.

Exclusion Criteria:

1. Diagnosable sleep disorder
2. Medication use or diagnosis of medical or psychiatric condition that may impact sleep/weight status
3. Current or planned treatment for weight control
4. Allergies or dietary restrictions that would prevent consumption of foods used in the study

Ages: 6 Years to 11 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 149 (Actual)
Dates: Start 2018-02-28 (Actual); Primary Completion 2023-03-01 (Actual); Study Completion 2023-09-19 (Actual)

PRIMARY OUTCOMES:
Change in BMIz | Change from baseline BMIz at 6 months
  change in body mass index z-score (accounting for child age and sex)

SECONDARY OUTCOMES:
Change in Body Composition | Change from baseline percent body fat at 6 months
  change in body composition (% body fat) will be estimated by air displacement plethysmography (BOD POD®; Life Measurement Instruments, Concord, CA)
Change in Waist Circumference | Change from baseline waist circumference at 6 months
  Change in measured waist circumference
Change in Insulin Resistance | Change from baseline HOMA-IR at 6 months
  Change in the homeostatic model assessment of insulin resistance (HOMA-IR)
Change in Blood Glucose Levels | Change from baseline blood glucose levels at 6 months
  2-hour blood glucose levels measured within the context of an oral glucose tolerance test
Change in Non-HDL cholesterol (non-HDL-C) | Change from baseline in Non-HDL-C at 6 months
  Total cholesterol (TC) minus HDL-C, includes LDL-C, VLDL-C, and atherogenic apo-B containing lipoproteins
Change in Insulin Sensitivity Index (ISI) | Change from baseline ISI at 6 months
  Insulin Sensitivity Index measured within the context of an oral glucose tolerance test
Change in Sleep Period | Change from baseline in the sleep period at 6 months
  Wrist-worn actigraphy
Change in Caloric Intake | Change from baseline in caloric intake at 6 months
  24-hr dietary recalls on two days used to estimate caloric intake
Change in Food Reinforcement | Change from baseline in food reinforcement at 6 months
  Measured using a validated computer activity (Behavioral Choice Task), which assesses motivation for a food reward
Change in Eating in the Absence of Hunger (EAH) | Change from baseline in EAH at 6 months
  Food consumed within the context of the eating in the absence of hunger paradigm
Change in Percent Time spent in Moderate to Vigorous Physical Activity (MVPA) | Change from baseline in MVPA at 6 months
  Waist-worn accelerometer

CONTACTS AND LOCATIONS:
Overall Officials: Chantelle N Hart, PhD, Principal Investigator — Temple University
Locations (1):
- Temple University, Philadelphia, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Spaeth AM, Hawley NL, Raynor HA, Jelalian E, Greer A, Crouter SE, Coffman DL, Carskadon MA, Owens JA, Wing RR, Hart CN. Sleep, energy balance, and meal timing in school-aged children. Sleep Med. 2019 Aug;60:139-144. doi: 10.1016/j.sleep.2019.02.003. Epub 2019 Feb 16. PMID 30905623